CLINICAL TRIAL: NCT04318860
Title: Postoperative Pain After Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/507-31
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Colorectal surgery; Numeric rating scale; Minimally invasive surgery; Risk factors
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate pain after elective colorectal surgery and to identify risk factors for postoperative pain.

Patients:All elective colorectal surgeries at the department of surgery, Umeå university Hospital, Umeå, Sweden from March 2013 to April 2017

Primary outcome:The primary outcome measurement is the numeric rating scale (NRS), graded from 0-10, on day of surgery, postoperative (POD) 1, 2, 3. The patients are questioned by nurses each morning on four postoperative days to score the maximum pain during the previous 24 hours using the NRS.

DETAILED DESCRIPTION:
This study aimed to quantify pain after elective colorectal surgery and to identify risk factors for postoperative pain.

Patients: This prospective cohort study includes all consecutive patients undergoing elective colorectal surgery at Umeå University Hospital in Sweden between March 2013 and April 2017.

Exclusion criteria: Patients who do not score pain at any of 4 postoperative days.

Primary outcome:The primary outcome measurement is the Numeric rating scale (NRS), graded from 0-10, where 0 = no pain and 10 = the worst imaginable pain [18]. Moderate pain is defined as NRS 4-6 and severe pain as NRS 7-10. The patients are questioned by nurses each morning after day of surgery, postoperative day. 1, postoperative day 2 and postoperative day 3 to score the maximum pain during the previous 24 hours using the NRS.

All data are registered in Enhanced recovery after surgery database (EISA)

Clinical variables: Baseline clinical variables are assessed preoperatively. They included age, gender, body mass index (BMI), smoking, a diabetes mellitus diagnosis and American Society of Anesthesia (ASA) class. The postoperative course is registered prospectively in Enhanced recovery after surgery register (EIAS) and include preoperative oncological treatment, a histopathologically verified cancer diagnosis, the length of hospital stay and complications, including any complication, Clavien-Dindo 3b or more and anastomotic leakage within 30 days after surgery High-sensitivity C-reactive protein (CRP) is measured every postoperative morning.

ELIGIBILITY:
Inclusion Criteria: Consecutive adults undergoing elective open and minimally invasive colorectal surgery at the Department of Surgery, Umeå University Hospital, from March 2013 to April 2017

Exclusion Criteria: Patients not scoring pain at any of 4 postoperative days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults undergoing elective colorectal surgery
Sampling Method: Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Maximum pain on day of surgery | Day of surgery
  Numeric rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain)
Maximum pain on postoperative day 1 | Postoperative day 1
  Numeric rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain)
Maximum pain on postoperative day 2 | Postoperative day 2
  Numeric rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain)
Maximum pain on postoperative day 3 | Postoperative day 3
  Numeric rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, prof, Principal Investigator — Dept Surgical and periopertive sciences, Umeå university, Sweden
Locations (1):
- Dept of Surgery, Inst of Surgical and Perioperative sciences, Umeå, Umea, Sweden